CLINICAL TRIAL: NCT02726152
Title: Randomised Control Trial: Polymer Clips Versus Endoloops for Closure of the Appendiceal Stump During Emergency Laparoscopic Appendicectomy (The PECAS Trial)
Brief Title: Polymer Clips Versus Endoloops for Closure of the Appendiceal Stump During Emergency Laparoscopic Appendicectomy
Acronym: PECAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Michael Wilson, Specialty Registrar, General Surgery, National Health Service, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015SA03
Record Dates: First submitted 2016-03-18; First posted 2016-04-01 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Appendicitis
Keywords: Diagnostic laparoscopy; Acute appendicitis; Appendiceal stump
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polymer clips (Experimental): Patients will be randomised to polymer clips for closure of the appendiceal stump
  Interventions: Procedure: Polymer clips for closure of the appendiceal stump
- Endoloops (Active Comparator): Patients will be randomised to endoloops for closure of the appendiceal stump
  Interventions: Procedure: Endoloops for closure of the appendiceal stump

INTERVENTIONS:
Procedure: Polymer clips for closure of the appendiceal stump — Application of polymer clips to the appendiceal stump
  Arms: Polymer clips
Procedure: Endoloops for closure of the appendiceal stump — Application of endoloops to the appendiceal stump
  Arms: Endoloops

SUMMARY:
The investigators propose a study to compare two methods of closing the stump of the appendix during an emergency excision of the appendix using a keyhole approach. One similarly designed study has been undertaken in another institution but there were not enough patients recruited to the study to allow meaningful conclusions to be drawn.

Any patient over the age of 16 years whom the investigators suspect to have acute appendicitis will be considered for recruitment to the study. During their exploratory keyhole surgery, if the surgical team feels that excision of the appendix is indicated then the patient will be randomly allocated to either polymer clips or endoloops to the part of the procedure where the stump (base) of the appendix is closed.

The main aim is to determine if polymer clips shorten the duration of the operation. The investigators will also determine if there is a difference between the rates of complications, the time spent in hospital and the number of times the participants had to be readmitted to hospital within 30 days.

DETAILED DESCRIPTION:
The investigators propose to perform a randomised control trial within NHS Tayside comparing two forms of appendiceal stump closure in emergency laparoscopic appendicectomy. A previous RCT examining this topic could have been better designed, with a small trial population and the absence of a power calculation.

All patients over 16 years old undergoing diagnostic laparoscopy for acute appendicitis will be eligible for recruitment to the trial and be consented prior to theatre. Intra-operatively, when the decision to perform an appendicectomy is taken, participants will be randomised to either the application of polymer (Locaclip) clips or endoloops to the appendiceal stump for closure during laparoscopic appendicectomy. The primary outcome will be operative time, while secondary outcomes include post-operative complications length of hospital stay and re-admission rate within 30 days. Participants will require no formal follow-up, either in the out-patient clinic or telephone consultations.

Statistical analysis will predominantly use Fisher's exact test to determine any statistically significant differences between each intervention arm, whilst group homogeneity will be analysed for other important patient parameters.

The investigators hypothesise that the operative time will be less in the polymer group compared to the endoloop group, while no significant difference will be seen in post-operative complications or other secondary outcomes between the two cohorts. The results of this RCT will add to the evidence-base for the use of polymer clips in appendiceal stump closure and potentially support its use for routine clinical practice. It is anticipated that it will take one year to recruit participants for the study and a further 30 days to complete follow up for the last participant recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspicion of acute appendicitis who are to do undergo diagnostic laparoscopy +/- appendicectomy
* Over the age of 16 years
* Able to give informed consent for inclusion in the study

Exclusion Criteria:

* Intraoperative decision to convert to open appendicectomy
* Primary open appendicectomy
* Under 16 years old
* Unable to give informed consent for participation in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative
  Is there difference in the overall operating time between the two cohorts

SECONDARY OUTCOMES:
Length of hospital stay (postoperative) | Up to 14 days
  Is there a significant difference in the length of postoperative stay between the two cohorts
Complications | 30 days
  Is there a difference in the rate of intraoperative and postoperative complications
Readmissions to hospital within 30 days of surgery | 30 days
  Is there a difference in the thirty day readmission rates between the two cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Ninewells Hospital, Dundee, Angus, United Kingdom

IPD SHARING:
Plan to Share IPD: No